CLINICAL TRIAL: NCT06120348
Title: Multi-center, Placebo-controlled, Randomized, Parallel Design, Superiority, Pivotal Clinical Trial to Evaluate the Efficacy and Safety of Application of Electrical Stimulation Around Eye After Laser Keratoplasty (LASEK) in Patients With Dry Eye Syndrome.
Brief Title: Study of Application of Pulse Electrical Stimulation Around Eye in Dry Eye Disease Patients Who Are Scheduled for Laser Epithelial Keratomileusis (LASEK) Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NE_DED_003
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Charge-Balanced, Symmetric Nerve Stimulation device 30 mins once a day for 4weeks(28days) and twice a week from the 5weeks to the 12 weeks.
  Interventions: Device: Charge-Balanced, Symmetric Nerve Stimulation
- Control Group (Sham Comparator): Sham device 30 mins once a day for 4weeks(28days) and twice a week from the 5weeks to the 12 weeks.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Charge-Balanced, Symmetric Nerve Stimulation — Charge-Balanced, Symmetric Nerve Stimulation device 30 mins once a day for 4weeks(28days) and twice a week from the 5weeks to the 12 weeks.
  Arms: Experimental Group
Device: Sham Stimulation — Sham device 30 mins once a day for 4weeks(28days) and twice a week from the 5weeks to the 12 weeks.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the efficacy and safety of applying pulse Electrical Stimulation around eye after laser keratoplasty (LASEK) in patients with dry eye syndrome.

DETAILED DESCRIPTION:
Duration of study period (per participant): Screening period (0-4weeks). Intervention period (12weeks).

Patient needs to visit site at least 8 times (Screening, baseline, 1 day, 3day, 1, 4, 8, 12weeks based on baseline). Baseline visit will be done on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 to 60
* Those who are scheduled to get LASEK surgery
* Those who have had dry eye symptoms for more than 3 months.
* According to the guidelines for diagnosing dry eye syndrome of Korean Corneal Disease Study Group, those who fall under Grade II or higher
* Those who TBUT test results of less than 10 seconds
* Those who OSDI score of 13 or higher
* Those who agreed to use contraception using a medically acceptable method during the period of clinical trial among Women of child bearing potential (WOCBP).
* A person who voluntarily agreed to participate in this clinical trial.

Exclusion Criteria:

* A person who has applied cyclosporin for the treatment of dry eye syndrome, drugs such as lipid-containing eye drops, topical steroid eye drops, IPL, etc., and medical devices for the treatment of dry eye syndrome within one month from the screening
* A person with an uncontrollable systemic chronic disease.
* Those who are allergic to drugs such as Fluorescein Solution or ophthalmic anesthetics
* In a case where there is a history of receiving ophthalmic surgery known to affect the tear layer within the last 6 months (e.g., Cataract, Punctal plug insertion, Pterygium surgery)
* A person who has eyelid diseases or structural abnormalities
* A person with acute eye infection or inflammation of the eyeball not related to Meibomian gland dysfunction
* A person with abnormalities in the eyelids or eyelashes
* A person with an eye condition or ophthalmic disease that is considered unsuitable for surgery
* A person who takes systemic drugs (e.g., tetracycline derivatives, antihistamine, isotretinoin)
* Pregnant or lactating women
* Those who can't understand or read the consent form of this clinical trial (e.g., illiterate or foreigners)
* Any other cases that PI considers hard to participate in this clinical trial (e.g., heart-related problems, seizure, epilepsy. Patients transplanted metal or electronic device in head & neck. Patient suffering from unknown pain. Patients who are warned not to use our clinical trial device or is prohibited from using it (e.g., pacemaker user).)
* Those who wore contact lenses within 72 hours before screening or who must wear contact lenses during the clinical trial period
* Those who have taken the relevant systemic drugs (steroids, immunosuppressants, omega-3 and anticholinergic drugs, etc.) within 30 days from the date of screening
* Those who are judged to have problems attaching electrodes due to inflammatory reactions or other dermatological problems in the skin around the orbit where the electrodes of medical devices are attached
* Those who participated in other clinical trial within 30 days from the screening date

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Tear break-up time (T-BUT) | baseline, 12 weeks
  Check the changes in Tear break-up time (T-BUT)
Changes in Visual Analogue Scale (VAS) score | baseline, 1 week
  Check the changes in Visual Analogue Scale (VAS) score

SECONDARY OUTCOMES:
Changes in Tear break-up time (T-BUT) | baseline, 1, 4, 8 weeks
  Check the changes in Tear break-up time (T-BUT)
Changes in 5-Item Dry Eye Questionnaire (DEQ-5) and Ocular Surface Disease Index (OSDI) score | baseline, 1, 4, 8, 12 weeks
  Check the changes in 5-Item Dry Eye Questionnaire Dry Eye Questionnaire (DEQ-5) and Ocular Surface Disease (OSDI) score
Changes in Visual Analogue Scale (VAS) score | baseline, 3 days, 4, 8, 12 weeks
  Check the changes in Visual Analogue Scale (VAS) score
Changes in Staining Score | baseline, 1, 4, 8, 12 weeks
  Check the changes in Staining Score
Changes in the length of the aesthesiometer's filament in centimeters | baseline, 1, 4, 8, 12 weeks
  Check the changes in the length of the aesthesiometer's filament in centimeters
Changes in Tear Volume | baseline, 1, 4, 8, 12 weeks
  Check the changes in Tear Volume

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hui Lim, Ph. D., MD, Principal Investigator — Department of Ophthalmology, Samsung Medical Center
Locations (6):
- South Korea (6):
  - HanGil Medical Foundation, Incheon
  - Department of Ophthalmology, Kangbuk Samsung Hospital, Seoul
  - Department of Ophthalmology, Severance Hospital, Seoul
  - Nune Eye Hospital, Seoul
  - Department of Ophthalmology, Samsung Medical Center, Seoul
  - Kim's Eye Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No